CLINICAL TRIAL: NCT06813430
Title: Enhancing Healing With Non-Contact Low-Frequency Ultrasound in Fingertip Amputation Treatment: A Prospective Comparative Cohort Study
Brief Title: Non-Contact Low-Frequency Ultrasound Vs Standard LaLonde Protocol for Fingertip Injury Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FY2025-115
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Non-contact Low Frequency Ultrasound; Lalonde Protocol; Fingertip Amputation
Keywords: non-contact low frequency ultrasound; Lalonde protocol; fingertip amputation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-Contact Low Frequency Ultrasound (Experimental): Lalonde therapy and non-contact low-frequency (UltraMIST) therapy - NCLF-US therapy involves delivering low-frequency (40 kHz), low-intensity (0.1-0.8 W/cm2) ultrasound energy via sterile water mist.
  Interventions: Device: Non-contact Low Frequency Ultrasound; Other: Lalonde Protocol (standard of care)
- Lalonde Protocol (Active Comparator): Standard of care local wound therapy using the Lalonde protocol - rinsing the site with clean water, applying a grease layer, wrapping with a one-inch gauze wrap, and securing with Coban tape.
  Interventions: Other: Lalonde Protocol (standard of care)

INTERVENTIONS:
Device: Non-contact Low Frequency Ultrasound — NCLF-US therapy involves delivering low-frequency (40 kHz), low-intensity (0.1-0.8 W/cm2) ultrasound energy via sterile water mist.
  Arms: Non-Contact Low Frequency Ultrasound
Other: Lalonde Protocol (standard of care) — Standard of care local wound therapy using the Lalonde protocol - rinsing the site with clean water, applying a grease layer, wrapping with a one-inch gauze wrap, and securing with Coban tape.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of non-contact low frequency ultrasound in populations sustaining fingertip amputations. The main question it aims to answer is:

• Does non-contact low frequency ultrasound significantly improve patient outcomes in patients sustaining acute fingertip amputations?

Researchers will compare non-contact low frequency ultrasound to a standard Lalonde protocol to answer this questions.

Participants will be randomized one of the two study arms and evaluated by wound care therapy. They will receive cohort appropriate therapy sessions 2-3 times per week with measurement of wound size once per week.

DETAILED DESCRIPTION:
Fingertip injuries rank among the most prevalent hand injuries, leading to nearly 5 million emergency department visits annually. Particularly common among adults, are lacerations, crush injuries, and avulsions affecting the thumb, index finger, and middle finger. As fingertip amputations encompass a diverse range of injuries involving soft tissue, bone, and/or nail, there is no singular recommended treatment as the standard of care. Instead, treatment is tailored to the individual patient, aiming to minimize pain, optimize healing, preserve sensory and motor function, and maintain an aesthetically acceptable appearance.

Possible treatment options for fingertip amputations without exposure of the distal phalanx include primary closure, healing by secondary intention, completion/revision amputation, full-thickness skin grafting, and split-thickness skin grafting, or flap coverage. However, when soft tissue allows, primary closure or healing by secondary intention have demonstrate positive and reliable outcomes.

New technologies, such as non-contact low-frequency ultrasound (NCLF-US), continue to be introduced to support healing of acute and chronic injuries to improve patient outcomes. While a moderate amount of research exists demonstrating safety and efficacy of NCLF-US in expediting the healing of chronic wounds, there is limited research on its efficacy in the treatment of acute injuries.

Given the significance of optimizing healing, especially in a population predominantly composed of young men engaged in manual labor, it is reasonable to wonder about the efficacy of NCLF-US in the treatment of fingertip amputations without exposed bone managed through secondary intention. This study aimed to compare the efficacy of NCLF-US in combination with standard treatment for secondary healing versus the standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older with an acute traumatic fingertip amputation without exposed bone or tendons (Allen 1, Tamai level 1; ICD-10 codes S68.5 and S68.6).

Exclusion Criteria:

* Patients less than 18 years old,
* Injuries involving exposed bone
* Those with diagnosis of vascular disease
* Individuals with clinical suspicion or diagnosis of infection
* Unable to comply with prescribed therapy sessions
* Patients undergoing primary closure or surgical intervention
* Patients experiencing subsequent trauma following treatment initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Wound Dimensions (mm2) | Assessed weekly. From date of randomization through study completion (an average of 8 weeks)
  Would dimensions will be measured in two dimensions using a ruler and recorded.
Time to Healing (days) | From randomization through study completion (an average of 8 weeks)
  Time to healing will be determined in days from randomization through study completion. This will vary between groups, but is expected to be complete by 8 weeks for all patients.

SECONDARY OUTCOMES:
Subjective Pain (Visual Analog Scale) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  The Visual Analog Scale, or VAS, will be used to measure subjective pain. Patients will report subjective pain on a scale of 1-10 with 10 indicating worse pain.
2 point discrimination (mm) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  Calipers will be used to determine patient 2-point discrimination status. A healthy patient is able to report discrimination between two points at 2-8mm at the fingertips. Larger values indicate worsening discrimination between two points and indicate worsening neurologic status.
Semmes Weinstein (Monofilament Sensitivity Test) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  A monofilament will be used to determine sensory status in the affected finger. Patients report yes or no when asked if they can sense the monofilament.
Grip Strength (lbs) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  A handgrip dynamometer will be used to determine the handgrip strength for patients in lbs. Larger numbers indicate increased strength.
Pinch Strength (lbs) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  A pinch dynamometer will be used to determine the pinch strength for patients in lbs. Larger numbers indicate increased strength.
Number of Visits (n) | From randomization through study completion (an average of 8 weeks)
  The number of visits the patient attends will be recorded. It is expected that patient enrollment in the study will be complete by an average of 8 weeks.
Functional Scores (Quick Disabilities of Arm, Shoulder, Hand) | Assessed weekly. From randomization through study completion (an average of 8 weeks)
  The Quick Disabilities of Arm, Shoulder, Hand (QuickDASH), a validating instrument, will be used to assess patient functional status. Scores range from 0-100. Higher scores indicate worse functional status.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In order to comply with the Health Insurance Portability and Accountability Act (HIPPA) as well as local/institutional regulations, only deidentified data can be provided from the primary investigator upon reasonable request. Independent review of the deidentified data to verify its accuracy will be permitted after article publication.

REFERENCES:
- [Background] Yao M, Hasturk H, Kantarci A, Gu G, Garcia-Lavin S, Fabbi M, Park N, Hayashi H, Attala K, French MA, Driver VR. A pilot study evaluating non-contact low-frequency ultrasound and underlying molecular mechanism on diabetic foot ulcers. Int Wound J. 2014 Dec;11(6):586-93. doi: 10.1111/iwj.12005. Epub 2012 Nov 19. PMID 23163982
- [Background] Kavros SJ, Schenck EC. Use of noncontact low-frequency ultrasound in the treatment of chronic foot and leg ulcerations: a 51-patient analysis. J Am Podiatr Med Assoc. 2007 Mar-Apr;97(2):95-101. doi: 10.7547/0970095. PMID 17369314
- [Background] Kavros SJ, Miller JL, Hanna SW. Treatment of ischemic wounds with noncontact, low-frequency ultrasound: the Mayo clinic experience, 2004-2006. Adv Skin Wound Care. 2007 Apr;20(4):221-6. doi: 10.1097/01.ASW.0000266660.88900.38. PMID 17415030
- [Background] Driver VR, Yao M, Miller CJ. Noncontact low-frequency ultrasound therapy in the treatment of chronic wounds: a meta-analysis. Wound Repair Regen. 2011 Jul-Aug;19(4):475-80. doi: 10.1111/j.1524-475X.2011.00701.x. Epub 2011 Jun 7. PMID 21649783
- [Background] Escandon J, Vivas AC, Perez R, Kirsner R, Davis S. A prospective pilot study of ultrasound therapy effectiveness in refractory venous leg ulcers. Int Wound J. 2012 Oct;9(5):570-8. doi: 10.1111/j.1742-481X.2011.00921.x. Epub 2012 Feb 1. PMID 22296347
- [Background] Olyaie M, Rad FS, Elahifar MA, Garkaz A, Mahsa G. High-frequency and noncontact low-frequency ultrasound therapy for venous leg ulcer treatment: a randomized, controlled study. Ostomy Wound Manage. 2013 Aug;59(8):14-20. PMID 23934374
- [Background] Kavros SJ, Liedl DA, Boon AJ, Miller JL, Hobbs JA, Andrews KL. Expedited wound healing with noncontact, low-frequency ultrasound therapy in chronic wounds: a retrospective analysis. Adv Skin Wound Care. 2008 Sep;21(9):416-23. doi: 10.1097/01.ASW.0000323546.04734.31. PMID 18769168
- [Background] Ennis WJ, Valdes W, Gainer M, Meneses P. Evaluation of clinical effectiveness of MIST ultrasound therapy for the healing of chronic wounds. Adv Skin Wound Care. 2006 Oct;19(8):437-46. doi: 10.1097/00129334-200610000-00011. PMID 17008814
- [Background] Ennis WJ, Foremann P, Mozen N, Massey J, Conner-Kerr T, Meneses P. Ultrasound therapy for recalcitrant diabetic foot ulcers: results of a randomized, double-blind, controlled, multicenter study. Ostomy Wound Manage. 2005 Aug;51(8):24-39. PMID 16234574
- [Background] Lee LP, Lau PY, Chan CW. A simple and efficient treatment for fingertip injuries. J Hand Surg Br. 1995 Feb;20(1):63-71. doi: 10.1016/s0266-7681(05)80019-1. PMID 7759939
- [Background] Mennen U, Wiese A. Fingertip injuries management with semi-occlusive dressing. J Hand Surg Br. 1993 Aug;18(4):416-22. doi: 10.1016/0266-7681(93)90139-7. PMID 8409649
- [Background] Lee DH, Mignemi ME, Crosby SN. Fingertip injuries: an update on management. J Am Acad Orthop Surg. 2013 Dec;21(12):756-66. doi: 10.5435/JAAOS-21-12-756. PMID 24292932
- [Background] Peterson SL, Peterson EL, Wheatley MJ. Management of fingertip amputations. J Hand Surg Am. 2014 Oct;39(10):2093-101. doi: 10.1016/j.jhsa.2014.04.025. PMID 25257490
- [Background] Sorock GS, Lombardi DA, Hauser RB, Eisen EA, Herrick RF, Mittleman MA. Acute traumatic occupational hand injuries: type, location, and severity. J Occup Environ Med. 2002 Apr;44(4):345-51. doi: 10.1097/00043764-200204000-00015. PMID 11977421